CLINICAL TRIAL: NCT04167163
Title: An Open-Label Phase 2 Study of Abaloparatide to Mitigate Distal Femoral Bone Loss Following Total Knee Arthroplasty
Brief Title: Abaloparatide Before Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Radius Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0685; A534255 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*G (Other: UW Madison); Protocol Version 3/22/2021 (Other: UW Madison)
Record Dates: First submitted 2019-10-29; First posted 2019-11-18 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Osteoporosis; Arthroplasties, Knee Replacement
MeSH Terms: conditions — Osteoporosis | interventions — abaloparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): Those with clinical osteoporosis who elect ABL treatment.
  ABL therapy will begin 3 months pre-TKA and continue for a total of 18 months. ABL will be administered by injection pen with dose of 80 mcg SC qDay.
  Interventions: Drug: Abaloparatide
- Comparator group (No Intervention): Those with clinical osteopenia who receive no treatment.

INTERVENTIONS:
Drug: Abaloparatide — 18 month ABL treatment
  Other Names: Tymlos
  Arms: Treatment group

SUMMARY:
The investigator hypothesizes that treating osteoporotic patients with abaloparatide prior to and after total knee arthroplasty will significantly reduce the amount of bone loss.

DETAILED DESCRIPTION:
In primary unilateral total knee arthroplasty patients, The investigator will examine the effect of daily abaloparatide therapy in clinical osteoporotic patients beginning 3 months pre-op and continued for a total of 15 months. This will be compared to osteopenic patients receiving no therapy as well as previously published values in untreated osteoporotic patients 12 months following Total Knee Arthroplasty (TKA).

ELIGIBILITY:
Inclusion Criteria

1. Post-menopausal women and men age ge ≥ 55 years and scheduled to undergo primary TKA at the University of Wisconsin Total Joint Program.
2. Osteoporosis, i.e., BMD T-score (using female reference data) ≤ -2.5 at the lumbar spine, femoral neck OR total hip or ≤ -1.1 with Vertebral Fracture Assessment confirmed vertebral fracture or history of low-trauma nonvertebral fracture in the past 5 years OR osteopenia, BMD T-score (using female reference data) -1.1 to -2.4 at the lumbar spine, femoral neck or total hip and no prior low-trauma fracture.
3. Serum calcium (albumin-corrected), serum creatinine and Parathyroid(PTH) values all within the normal range and 25(OH)D > 10 ng/mL.
4. Willing to supplement with daily calcium and/or vitamin D3 at protocol specified doses.
5. Able to provide written informed consent.

Exclusion Criteria

1. Unevaluable distal femur BMD due to hardware or other artifacts.
2. History of bone disorders (e.g., Paget's disease) other than osteoporosis.
3. History of prior external beam or implant radiation therapy involving the skeleton other than radioiodine.
4. History of chronic or recurrent renal, hepatic, pulmonary, allergic, cardiovascular, gastrointestinal, endocrine, central nervous system, hematologic or metabolic diseases, or immunologic, emotional and/or psychiatric disturbances that, in opinion of the principal investigator, would compromise study data validity.
5. History of Cushing's disease, growth hormone deficiency or excess, hyperthyroidism, hypo- or hyperparathyroidism or malabsorptive syndromes within the past year.
6. History of significantly impaired renal function (serum creatinine >2.0 mg/dL. If the serum creatinine is > 1.5 and ≤ 2.0 mg/dL, the calculated creatinine clearance (Cockcroft-Gault) must be ≥ 37 mL/min.
7. History of nephrolithiasis or urolithiasis within the past five years.
8. History of cancer in prior 5 years (basal cell or squamous skin cancer is permissible).
9. History of osteosarcoma at any time.
10. Patients known to be positive for Hepatitis B, Hepatitis C, HIV-1 or HIV-2.
11. Known hypersensitivity to any of the test materials or related compounds.
12. Prior treatment with PTH- or PTHrP-derived drugs, (ABL, teriparatide or PTH (1-84)).
13. Prior treatment with intravenous bisphosphonates at any time or oral bisphosphonates within the past three years. Patients who had received a short course of oral bisphosphonate therapy (3 months or less) may be enrolled as long as the treatment occurred 6 or more months prior to enrollment.
14. Treatment with fluoride or strontium in the past five years or prior treatment with bone-acting investigational agents at any time.
15. Treatment with calcitonin the past 6 months or denosumab in the past 18 months.
16. Treatment with anticonvulsants affecting vitamin D metabolism (phenobarbital, phenytoin, carbamazepine or primidone) or chronic heparin within the prior 6 months.
17. Treatment with anabolic steroids or calcineurin inhibitors (cyclosporin, tacrolimus)
18. Daily treatment with oral, intranasal or inhaled glucocorticoids in the prior 12 months.
19. Exposure to any investigational drug within 12 months.
20. Consumption of > 2 alcoholic drinks per day or use of illegal drugs within 12 months of screening.
21. Not suitable for study participation due to other reasons at the investigators discretion.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Change in Distal femoral Bone mineral density (BMD) at the 25% regions of interest (ROIs) | Baseline and 18 months
  Bone mineral density change at the 25% ROI of the surgical leg

SECONDARY OUTCOMES:
Change in Distal femoral BMD at the 15% and 60 %ROI | Baseline and 18 months
  Bone mineral density change at the 15% and 60% ROI of the surgical leg
Change in Femur cortical thickness at the 15%, 25% and 60% femur ROIs | Baseline and 18 months
  Cortical thickness change at the 15% and 60% ROI of the surgical leg
TBS assessment by TRIP at the 15%, 25% and 60% femur ROIs | 18 months
  Trabecular bone score (TBS) assessment by Texture Research Investigation (Platform (TRIP) software change at the 15%, 25% and 60% femur ROIs (TBS >1.350 is normal; TBS between 1.200 and 1.350 is indicative of partially degraded microarchitecture; and TBS<1.200 equals degraded microarchitecture)
Knee injury & Osteoarthritis Outcome Score (KOOS) JR | 18 months
  Patient reported knee function score. The KOOS, JR was developed from the original long version of the Knee injury and Osteoarthritis Outcome Score (KOOS) survey using Rasch analysis. The KOOS, JR contains 7 items from the original KOOS survey. Items are coded from 0 to 4, none to extreme respectively. KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score (0-100). The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Change in Veterans RAND 12 (VR-12) Question Health Survey score | Baseline and 18 months
  12 Item Health Survey using patient's self assessment of their perspective of their health and ability to do daily functions. Scores are derived using an algorithm that is referenced to a metric centered at 50.0 where a zero score indicates the lowest level of health and 100 indicates the highest level of health.
Forgotten Joint Survey(FJS) score | 18 months
  FJS-12 consists of 12 questions and is scored using a 5-point response format with the raw scores transformed onto a 0- to 100-point scale.
  High scores indicate good outcome, that is, a high degree of forgetting the joint in everyday life (forgotten joint phenomenon).
Change in body composition using bioelectrical impedance analysis of lean mass | Baseline and 18 months
  Change in body composition using bioelectrical impedance analysis of lean mass.
Change in body composition using bioelectrical impedance analysis of skeletal mass. | Baseline and 18 months
  Change in body composition using bioelectrical impedance analysis of skeletal mass.
Change in body composition using bioelectrical impedance analysis of fat mass. | Baseline and 18 months
  Change in body composition using bioelectrical impedance analysis of fat mass.
TKA complications: Number of participants needed revision surgery | 18 months
  TKA complications: Number of participants needed revision surgery
TKA complications: Number of participants had fracture | 18 months
  TKA complications: Number of participants had fracture
Precision Error on Knee Bone Density Measurement | up to 15 months
  Precision assessment in the field of bone densitometry is the process whereby the ability of the instrument and the technologist to reproduce similar results, given no real biologic change, is tested. The mathematical result of precision assessment is called the precision error. To achieve statistical power, the investigators will take duplicate knee bone density measurements on 30 participants at either their 6 month or 15 month visit. The standard deviation for each participant is calculated, then the root mean square standard deviation for the group is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Binkley, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maradit Kremers H, Larson DR, Crowson CS, Kremers WK, Washington RE, Steiner CA, Jiranek WA, Berry DJ. Prevalence of Total Hip and Knee Replacement in the United States. J Bone Joint Surg Am. 2015 Sep 2;97(17):1386-97. doi: 10.2106/JBJS.N.01141. PMID 26333733
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Chang CB, Kim TK, Kang YG, Seong SC, Kang SB. Prevalence of osteoporosis in female patients with advanced knee osteoarthritis undergoing total knee arthroplasty. J Korean Med Sci. 2014 Oct;29(10):1425-31. doi: 10.3346/jkms.2014.29.10.1425. Epub 2014 Oct 8. PMID 25368498
- [Background] Lingard EA, Mitchell SY, Francis RM, Rawlings D, Peaston R, Birrell FN, McCaskie AW. The prevalence of osteoporosis in patients with severe hip and knee osteoarthritis awaiting joint arthroplasty. Age Ageing. 2010 Mar;39(2):234-9. doi: 10.1093/ageing/afp222. Epub 2009 Dec 23. PMID 20032523
- [Background] Frenzel S, Vecsei V, Negrin L. Periprosthetic femoral fractures--incidence, classification problems and the proposal of a modified classification scheme. Int Orthop. 2015 Oct;39(10):1909-20. doi: 10.1007/s00264-015-2967-4. Epub 2015 Sep 2. PMID 26330085
- [Background] Sarmah SS, Patel S, Reading G, El-Husseiny M, Douglas S, Haddad FS. Periprosthetic fractures around total knee arthroplasty. Ann R Coll Surg Engl. 2012 Jul;94(5):302-7. doi: 10.1308/003588412X13171221592537. PMID 22943223
- [Background] Della Rocca GJ, Leung KS, Pape HC. Periprosthetic fractures: epidemiology and future projections. J Orthop Trauma. 2011 Jun;25 Suppl 2:S66-70. doi: 10.1097/BOT.0b013e31821b8c28. PMID 21566478
- [Background] Head J 2017 Periprosthetic distal femur fractures: Review of current treatment options. Reconstructive Review 7:NO4
- [Background] Meek RM, Norwood T, Smith R, Brenkel IJ, Howie CR. The risk of peri-prosthetic fracture after primary and revision total hip and knee replacement. J Bone Joint Surg Br. 2011 Jan;93(1):96-101. doi: 10.1302/0301-620X.93B1.25087. PMID 21196551
- [Background] Hoffmann MF, Jones CB, Sietsema DL, Koenig SJ, Tornetta P 3rd. Outcome of periprosthetic distal femoral fractures following knee arthroplasty. Injury. 2012 Jul;43(7):1084-9. doi: 10.1016/j.injury.2012.01.025. Epub 2012 Feb 18. PMID 22348954
- [Background] Reeves RA, Schairer WW, Jevsevar DS. Costs and Risk Factors for Hospital Readmission After Periprosthetic Knee Fractures in the United States. J Arthroplasty. 2018 Feb;33(2):324-330.e1. doi: 10.1016/j.arth.2017.09.024. Epub 2017 Sep 23. PMID 29066112
- [Background] Lizaur-Utrilla A, Miralles-Munoz FA, Sanz-Reig J. Functional outcome of total knee arthroplasty after periprosthetic distal femoral fracture. J Arthroplasty. 2013 Oct;28(9):1585-8. doi: 10.1016/j.arth.2013.03.007. Epub 2013 Apr 17. PMID 23602235
- [Background] Ruder JA, Hart GP, Kneisl JS, Springer BD, Karunakar MA. Predictors of Functional Recovery Following Periprosthetic Distal Femur Fractures. J Arthroplasty. 2017 May;32(5):1571-1575. doi: 10.1016/j.arth.2016.12.013. Epub 2016 Dec 23. PMID 28131543
- [Background] Gazdzik TS, Gajda T, Kaleta M. Bone mineral density changes after total knee arthroplasty: one-year follow-up. J Clin Densitom. 2008 Jul-Sep;11(3):345-50. doi: 10.1016/j.jocd.2008.04.007. Epub 2008 Jul 10. PMID 18619880
- [Background] Windisch C, Windisch B, Kolb W, Kolb K, Grutzner P, Roth A. Osteodensitometry measurements of periprosthetic bone using dual energy X-ray absorptiometry following total knee arthroplasty. Arch Orthop Trauma Surg. 2012 Nov;132(11):1595-601. doi: 10.1007/s00402-012-1601-9. Epub 2012 Aug 12. PMID 22886240
- [Background] Soininvaara TA, Miettinen HJ, Jurvelin JS, Suomalainen OT, Alhava EM, Kroger HP. Periprosthetic femoral bone loss after total knee arthroplasty: 1-year follow-up study of 69 patients. Knee. 2004 Aug;11(4):297-302. doi: 10.1016/j.knee.2003.09.006. PMID 15261216
- [Background] Minoda Y, Ikebuchi M, Kobayashi A, Iwaki H, Inori F, Nakamura H. A cemented mobile-bearing total knee replacement prevents periprosthetic loss of bone mineral density around the femoral component: a matched cohort study. J Bone Joint Surg Br. 2010 Jun;92(6):794-8. doi: 10.1302/0301-620X.92B6.23159. PMID 20513875
- [Background] Jaroma A, Soininvaara T, Kroger H. Periprosthetic tibial bone mineral density changes after total knee arthroplasty. Acta Orthop. 2016 Jun;87(3):268-73. doi: 10.3109/17453674.2016.1173982. Epub 2016 Apr 27. PMID 27120266
- [Background] Au AG, James Raso V, Liggins AB, Amirfazli A. Contribution of loading conditions and material properties to stress shielding near the tibial component of total knee replacements. J Biomech. 2007;40(6):1410-6. doi: 10.1016/j.jbiomech.2006.05.020. Epub 2006 Jul 17. PMID 16846605
- [Background] Moon YW, Kim HJ, Ahn HS, Lee DH. Serial Changes of Quadriceps and Hamstring Muscle Strength Following Total Knee Arthroplasty: A Meta-Analysis. PLoS One. 2016 Feb 5;11(2):e0148193. doi: 10.1371/journal.pone.0148193. eCollection 2016. PMID 26849808
- [Background] Stevens JE, Mizner RL, Snyder-Mackler L. Quadriceps strength and volitional activation before and after total knee arthroplasty for osteoarthritis. J Orthop Res. 2003 Sep;21(5):775-9. doi: 10.1016/S0736-0266(03)00052-4. PMID 12919862
- [Background] Thomas B, Binkley N, Anderson PA, Krueger D. DXA Measured Distal Femur Bone Mineral Density in Patients After Total Knee Arthroplasty: Method Development and Reproducibility. J Clin Densitom. 2019 Jan-Mar;22(1):67-73. doi: 10.1016/j.jocd.2018.08.003. Epub 2018 Aug 13. PMID 30228047
- [Background] Blaty T, Krueger D, Illgen R, Squire M, Heiderscheit B, Binkley N, Anderson P. DXA evaluation of femoral bone mineral density and cortical width in patients with prior total knee arthroplasty. Osteoporos Int. 2019 Feb;30(2):383-390. doi: 10.1007/s00198-018-4682-7. Epub 2018 Aug 31. PMID 30171301
- [Background] Soininvaara T, Kroger H, Jurvelin JS, Miettinen H, Suomalainen O, Alhava E. Measurement of bone density around total knee arthroplasty using fan-beam dual energy X-ray absorptiometry. Calcif Tissue Int. 2000 Sep;67(3):267-72. doi: 10.1007/s002230001111. PMID 10954783
- [Background] Jaroma AV, Soininvaara TA, Kroger H. Effect of one-year post-operative alendronate treatment on periprosthetic bone after total knee arthroplasty. A seven-year randomised controlled trial of 26 patients. Bone Joint J. 2015 Mar;97-B(3):337-45. doi: 10.1302/0301-620X.97B3.33643. PMID 25737517
- [Background] Suzuki T, Sukezaki F, Shibuki T, Toyoshima Y, Nagai T, Inagaki K. Teriparatide Administration Increases Periprosthetic Bone Mineral Density After Total Knee Arthroplasty: A Prospective Study. J Arthroplasty. 2018 Jan;33(1):79-85. doi: 10.1016/j.arth.2017.07.026. Epub 2017 Jul 25. PMID 28869116
- [Background] Kaneko T, Otani T, Kono N, Mochizuki Y, Mori T, Nango N, Ikegami H, Musha Y. Weekly injection of teriparatide for bone ingrowth after cementless total knee arthroplasty. J Orthop Surg (Hong Kong). 2016 Apr;24(1):16-21. doi: 10.1177/230949901602400106. PMID 27122506
- [Background] Kobayashi N, Inaba Y, Uchiyama M, Ike H, Kubota S, Saito T. Teriparatide Versus Alendronate for the Preservation of Bone Mineral Density After Total Hip Arthroplasty - A randomized Controlled Trial. J Arthroplasty. 2016 Jan;31(1):333-8. doi: 10.1016/j.arth.2015.07.017. Epub 2015 Jul 17. PMID 26260784
- [Background] Teng S, Yi C, Krettek C, Jagodzinski M. Bisphosphonate Use and Risk of Implant Revision after Total Hip/Knee Arthroplasty: A Meta-Analysis of Observational Studies. PLoS One. 2015 Oct 7;10(10):e0139927. doi: 10.1371/journal.pone.0139927. eCollection 2015. PMID 26444555
- [Background] Smee DJ, Anson JM, Waddington GS, Berry HL. Association between Physical Functionality and Falls Risk in Community-Living Older Adults. Curr Gerontol Geriatr Res. 2012;2012:864516. doi: 10.1155/2012/864516. Epub 2012 Dec 4. PMID 23304137
- [Background] Binkley N, Krueger D, Buehring B. What's in a name revisited: should osteoporosis and sarcopenia be considered components of "dysmobility syndrome?". Osteoporos Int. 2013 Dec;24(12):2955-9. doi: 10.1007/s00198-013-2427-1. Epub 2013 Aug 1. PMID 23903951
- [Background] Buehring B, Hansen KE, Lewis BL, Cummings SR, Lane NE, Binkley N, Ensrud KE, Cawthon PM; Osteoporotic Fractures in Men (MrOS) Study Research Group. Dysmobility Syndrome Independently Increases Fracture Risk in the Osteoporotic Fractures in Men (MrOS) Prospective Cohort Study. J Bone Miner Res. 2018 Sep;33(9):1622-1629. doi: 10.1002/jbmr.3455. Epub 2018 Jun 21. PMID 29701911
- [Background] Meier W, Mizner RL, Marcus RL, Dibble LE, Peters C, Lastayo PC. Total knee arthroplasty: muscle impairments, functional limitations, and recommended rehabilitation approaches. J Orthop Sports Phys Ther. 2008 May;38(5):246-56. doi: 10.2519/jospt.2008.2715. Epub 2007 Dec 14. PMID 18448878
- [Background] Valtonen A, Poyhonen T, Heinonen A, Sipila S. Muscle deficits persist after unilateral knee replacement and have implications for rehabilitation. Phys Ther. 2009 Oct;89(10):1072-9. doi: 10.2522/ptj.20070295. Epub 2009 Aug 27. PMID 19713269
- [Background] Mizner RL, Petterson SC, Stevens JE, Vandenborne K, Snyder-Mackler L. Early quadriceps strength loss after total knee arthroplasty. The contributions of muscle atrophy and failure of voluntary muscle activation. J Bone Joint Surg Am. 2005 May;87(5):1047-53. doi: 10.2106/JBJS.D.01992. PMID 15866968
- [Background] Yamada Y, Schoeller DA, Nakamura E, Morimoto T, Kimura M, Oda S. Extracellular water may mask actual muscle atrophy during aging. J Gerontol A Biol Sci Med Sci. 2010 May;65(5):510-6. doi: 10.1093/gerona/glq001. Epub 2010 Feb 4. PMID 20133393
- [Background] Buehring B, Siglinsky E, Krueger D, Evans W, Hellerstein M, Yamada Y, Binkley N. Comparison of muscle/lean mass measurement methods: correlation with functional and biochemical testing. Osteoporos Int. 2018 Mar;29(3):675-683. doi: 10.1007/s00198-017-4315-6. Epub 2017 Dec 2. PMID 29198074
- [Background] Liu Y, Levack AE, Marty E, Or O, Samuels BP, Redko M, Lane JM. Anabolic agents: what is beyond osteoporosis? Osteoporos Int. 2018 May;29(5):1009-1022. doi: 10.1007/s00198-018-4507-8. Epub 2018 Apr 7. PMID 29627891
- [Background] Prince JM, Bernatz JT, Binkley N, Abdel MP, Anderson PA. Changes in femoral bone mineral density after total knee arthroplasty: a systematic review and meta-analysis. Arch Osteoporos. 2019 Feb 23;14(1):23. doi: 10.1007/s11657-019-0572-7. PMID 30798359
- [Background] Bernatz JT, Brooks AE, Squire MW, Illgen RI 2nd, Binkley NC, Anderson PA. Osteoporosis Is Common and Undertreated Prior to Total Joint Arthroplasty. J Arthroplasty. 2019 Jul;34(7):1347-1353. doi: 10.1016/j.arth.2019.03.044. Epub 2019 Mar 28. PMID 30992237
- [Background] Bernatz JT, Krueger DC, Squire MW, Illgen RL 2nd, Binkley NC, Anderson PA. Unrecognized Osteoporosis Is Common in Patients With a Well-Functioning Total Knee Arthroplasty. J Arthroplasty. 2019 Oct;34(10):2347-2350. doi: 10.1016/j.arth.2019.05.041. Epub 2019 May 30. PMID 31227302
- [Background] Yamada Y, Masuo Y, Yokoyama K, Hashii Y, Ando S, Okayama Y, Morimoto T, Kimura M, Oda S. Proximal electrode placement improves the estimation of body composition in obese and lean elderly during segmental bioelectrical impedance analysis. Eur J Appl Physiol. 2009 Sep;107(2):135-44. doi: 10.1007/s00421-009-1106-6. Epub 2009 Jun 17. PMID 19533166
- [Background] Miller PD, Hattersley G, Riis BJ, Williams GC, Lau E, Russo LA, Alexandersen P, Zerbini CA, Hu MY, Harris AG, Fitzpatrick LA, Cosman F, Christiansen C; ACTIVE Study Investigators. Effect of Abaloparatide vs Placebo on New Vertebral Fractures in Postmenopausal Women With Osteoporosis: A Randomized Clinical Trial. JAMA. 2016 Aug 16;316(7):722-33. doi: 10.1001/jama.2016.11136. PMID 27533157